CLINICAL TRIAL: NCT00624793
Title: Acupuncture for Chronic Nausea in HIV: A Randomized Clinical Trial
Brief Title: Acupuncture for Nausea in HIV
Acronym: AcuN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-0339
Record Dates: First submitted 2008-02-19; First posted 2008-02-27 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections
Keywords: Nausea; Vomiting; Retching; HIV/AIDS; Symptom Management; Complementary Therapies
MeSH Terms: conditions — HIV Infections; Nausea; Vomiting; Acquired Immunodeficiency Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- I. Standard (Experimental): Standard - Formula Acup Protocol
  Interventions: Other: Acupuncture
- 2. Individualized (Experimental): Individualized Acup protocol based on TCM diagnosis
  Interventions: Other: Individualized Acup based on TCM diagnosis
- 3 (Sham Comparator): (Control Group) Sham acupuncture
  Interventions: Other: Sham Acup

INTERVENTIONS:
Other: Acupuncture — Standard Acup point protocol for treating nausea
  Arms: I. Standard
Other: Individualized Acup based on TCM diagnosis — Acup
  Arms: 2. Individualized
Other: Sham Acup — Sham Acup - Non-Active
  Arms: 3

SUMMARY:
The subjects in this research study will be 159 men and women with HIV infection who have a history of chronic nausea for three months or greater and show evidence of two or more episodes of nausea and/or report a duration of two hours or more (per day) in baseline symptom diaries. Subjects will be randomized (by chance) to one of three conditions: Condition 1, subjects receive Standard acupuncture (active treatment); Condition 2, subjects receive Individualized acupuncture based on Traditional Chinese Medical Diagnosis (active treatment); Condition 3, (Control Group), subjects receive Sham acupuncture. Subjects in Conditions 1, 2, & 3 will attend scheduled sessions over 24 weeks.

DETAILED DESCRIPTION:
The subjects in the proposed experiment will be 159 men and women with HIV infection who have a history of chronic nausea for three months or greater and show evidence of two or more episodes of nausea and/or report a duration of 2 hours or greater (per day) in prospective baseline symptom diaries. Subjects will be randomized to one of three experimental intervention conditions: Condition 1, subjects receive Standard acupuncture; Condition 2, subjects receive Individualized acupuncture based on Traditional Chinese Medical Diagnosis; Condition 3, (Control Group), subjects receive Sham acupuncture. Subjects in Conditions 1, 2, & 3 will attend 16 scheduled sessions over 24 weeks. All subjects will: be assessed by a diagnostic acupuncturist (blinded to treatment assignments); be administered the same instruments; and submit their symptom diaries for data entry and analysis. After a screening/intake session, randomization and treatment sessions will follow. There will be four weeks of twice weekly treatment sessions, four weekly treatment sessions and three follow-up sessions. All conditions will be identical in duration and be administered by licensed acupuncturists trained in Traditional Chinese Medicine. This study is a prospective, randomized, controlled, blinded (subject and evaluator), parallel groups clinical trial aimed at reducing chronic nausea and improving quality of life in persons with HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women HIV positive or CDC AIDS diagnosed
* History of chronic nausea for three months or greater
* Experience an average of two or more episodes of nausea and/or who experience an average duration of 2 hours or more (of nausea) per day
* Verification from Primary provider of subject's: HIV status, knowledge of patient's nausea and their agreement that their patient is clinically suitable for the study.
* Individuals able to successfully complete a mini-mental status exam
* Individuals who understand and agree to complete daily symptom diaries for the duration of the study.
* Individuals taking antiretroviral combinations must have completed an initial 8 weeks of a stable regime (same drug(s), dose & frequency) prior to entry into the study.
* Individuals taking anti-emetic medications must be on a stable regime (same drug, dose & frequency) for at least fourteen days prior to entry into the study.
* Individuals on all other medications which may have nausea listed as a side effect must be on a stable regime (same drug(s), dose & frequency) for at least fourteen (14) days prior to entry in the study

Exclusion Criteria:

* Individuals with an acute medical condition, i.e. pneumocystis carinii pneumonia, tuberculosis and or other opportunistic infections or conditions that would require medical attention.
* Pregnant women
* Individuals receiving acupuncture currently and less than 6 months prior to enrollment.
* Individuals currently receiving other types of complementary therapies such as herbs, massage, acupressure wrist bands, reiki etc.
* Individuals with plans for travel, lifestyle change, or other activity that would preclude attending all of the planned study sessions and/or recording daily diary information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2005-05; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
INVR - symptom diary Clinical Global Impression Scales | Baseline, treatment and follow-ups sessions

SECONDARY OUTCOMES:
QOL scale MOS-SF-36 subscales | Baseline, treatment and follow-up session

CONTACTS AND LOCATIONS:
Overall Officials: Joyce K Anastasi, PhD, Principal Investigator — New York University